CLINICAL TRIAL: NCT03111186
Title: A Randomized Trial Comparing Ibuprofen Plus Acetaminophen Versus Oxycodone Alone After Outpatient Soft Tissue Hand Surgery
Brief Title: Ibuprofen Plus Acetaminophen Versus Oxycodone Alone After Hand Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Alidad Ghiassi, Assistant Professor of Clinical Orthopaedic Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS-15-00706
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-06

CONDITIONS: Carpal Tunnel Syndrome; Dupuytren Contracture; Trigger Digit; Ganglion Cysts; De Quervain Disease
Keywords: oxycodone; ibuprofen; acetaminophen; soft-tissue hand surgery; carpal tunnel release; Dupuytren contracture release; Trigger digit release; Ganglion cyst removal; De Quervain's release
MeSH Terms: conditions — Carpal Tunnel Syndrome; Dupuytren Contracture; Trigger Finger Disorder; Ganglion Cysts; De Quervain Disease | interventions — Oxycodone; Ibuprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Patients of either sex, greater than 18 years of age, scheduled to undergo elective outpatient soft tissue hand surgery for one of the following procedures: carpal tunnel release, Dupuytren contracture release, trigger digit release, ganglion cyst removal, De Quervain's release, whose primary language is English or Spanish
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Opiate group (Active Comparator): Group receiving oxycodone alone (oxycodone HCl 5 mg up to six times daily as needed for pain)
  Interventions: Drug: Oxycodone Hcl 5Mg
- Non-opiate group (Active Comparator): Group receiving ibuprofen and acetaminophen (acetaminophen 650 mg up to four times daily and ibuprofen 400 mg up to six times daily as need for pain)
  Interventions: Drug: Ibuprofen 400 mg; Drug: Acetaminophen 650 mg

INTERVENTIONS:
Drug: Oxycodone Hcl 5Mg — oxycodone HCl 5 mg up to six times daily as needed for pain
  Other Names: oxycodone
  Arms: Opiate group
Drug: Ibuprofen 400 mg — Ibuprofen 400 mg up to six times daily as needed for pain
  Arms: Non-opiate group
Drug: Acetaminophen 650 mg — Acetaminophen 650 mg up to four times daily as needed for pain
  Arms: Non-opiate group

SUMMARY:
This study is about pain control and medication following outpatient soft-tissue hand surgery. We hope to learn if ibuprofen and acetaminophen will achieve similar pain relief and satisfaction when compared with oxycodone alone.

DETAILED DESCRIPTION:
Opiate analgesics remain the most popular option following outpatient hand surgery despite growing evidence that non-opiate analgesics may provide equivalent pain relief with fewer adverse effects and greater overall satisfaction. The purpose of this randomized trial is to compare the efficacy, side effect profiles and satisfaction associated with Ibuprofen plus Acetaminophen versus Oxycodone alone following outpatient hand surgery. No previous studies have compared the use of opiate analgesics with acetaminophen/ibuprofen following outpatient hand surgery. Patients will be randomized to receive either oxycodone alone or acetaminophen and ibuprofen following outpatient soft tissue hand surgery. Patients will be randomized to receive one of the two aforementioned pain regimens. Patients will be given a booklet in which to record pain level by visual analog scale (VAS), satisfaction with pain control, brief pain inventory and any side effects. Patients will be seen in clinic 1 week after surgery to review symptoms. Patients may also be contacted by phone to review daily log of symptoms. Patients will be seen in clinic 1 week after surgery per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* scheduled to undergo elective outpatient soft tissue hand surgery for one of the following procedures: Carpal tunnel release, Dupuytren contracture release, trigger digit release, ganglion cyst removal, de Quervain's release.
* primary language is English or Spanish

Exclusion Criteria:

* any pre-existing condition requiring preoperative opiate analgesia, eg chronic pain syndrome
* allergy to acetaminophen, ibuprofen, or oxycodone
* renal impairment or liver disease either documented based on history or when preoperative creatinine, BUN, or liver function tests are outside the normal range provided by the lab
* peptic ulcer disease or any history of gastrointestinal bleeding
* coagulopathy documented on history, review of systems, or based on preoperative lab testing where PT, PTT, or INR are outside the normal range provided by the lab
* pregnancy based on positive beta-HCG test which is performed on the day of the surgical procedure as is standard protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
change in VAS pain scale | baseline, daily - up to 1 week postoperative
  Visual Analog Score - pain scale, patient questionnaire

SECONDARY OUTCOMES:
change in Brief Pain Index | baseline, daily - up to 1 week postoperative
  Brief Pain Index - pain scale, patient questionnaire
change in pain diary | baseline, daily - up to 1 week postoperative
  Pain Diary - pain scale, patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alidad Ghiassi, MD, Principal Investigator — University of Southern California
Locations (1):
- Keck School of Medicine of the University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as required with the USC Health Sciences Institutional Review Board. Participant data will be coded with coding identifiers kept separately by research personnel only and destroyed upon completion of the study.

REFERENCES:
- [Background] Coluzzi F, Bragazzi L, Di Bussolo E, Pizza G, Mattia C. Determinants of patient satisfaction in postoperative pain management following hand ambulatory day-surgery. Minerva Med. 2011 Jun;102(3):177-86. PMID 21593720
- [Background] Munns JJ, Awan HM. Trends in carpal tunnel surgery: an online survey of members of the American Society for Surgery of the Hand. J Hand Surg Am. 2015 Apr;40(4):767-71.e2. doi: 10.1016/j.jhsa.2014.12.046. Epub 2015 Mar 4. PMID 25747738
- [Background] Manchikanti L, Singh A. Therapeutic opioids: a ten-year perspective on the complexities and complications of the escalating use, abuse, and nonmedical use of opioids. Pain Physician. 2008 Mar;11(2 Suppl):S63-88. PMID 18443641
- [Background] Rodgers J, Cunningham K, Fitzgerald K, Finnerty E. Opioid consumption following outpatient upper extremity surgery. J Hand Surg Am. 2012 Apr;37(4):645-50. doi: 10.1016/j.jhsa.2012.01.035. Epub 2012 Mar 10. PMID 22410178
- [Background] Nauta M, Landsmeer ML, Koren G. Codeine-acetaminophen versus nonsteroidal anti-inflammatory drugs in the treatment of post-abdominal surgery pain: a systematic review of randomized trials. Am J Surg. 2009 Aug;198(2):256-61. doi: 10.1016/j.amjsurg.2008.11.044. PMID 19628064
- [Background] Rawal N, Allvin R, Amilon A, Ohlsson T, Hallen J. Postoperative analgesia at home after ambulatory hand surgery: a controlled comparison of tramadol, metamizol, and paracetamol. Anesth Analg. 2001 Feb;92(2):347-51. doi: 10.1097/00000539-200102000-00013. PMID 11159230
- [Background] Mitchell A, van Zanten SV, Inglis K, Porter G. A randomized controlled trial comparing acetaminophen plus ibuprofen versus acetaminophen plus codeine plus caffeine after outpatient general surgery. J Am Coll Surg. 2008 Mar;206(3):472-9. doi: 10.1016/j.jamcollsurg.2007.09.006. Epub 2007 Nov 26. PMID 18308218
- [Background] Joris J. Efficacy of nonsteroidal antiinflammatory drugs in postoperative pain. Acta Anaesthesiol Belg. 1996;47(3):115-23. PMID 8959196
- [Background] Ong CK, Seymour RA, Lirk P, Merry AF. Combining paracetamol (acetaminophen) with nonsteroidal antiinflammatory drugs: a qualitative systematic review of analgesic efficacy for acute postoperative pain. Anesth Analg. 2010 Apr 1;110(4):1170-9. doi: 10.1213/ANE.0b013e3181cf9281. Epub 2010 Feb 8. PMID 20142348
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Background] McCartney CJ, Brull R, Chan VW, Katz J, Abbas S, Graham B, Nova H, Rawson R, Anastakis DJ, von Schroeder H. Early but no long-term benefit of regional compared with general anesthesia for ambulatory hand surgery. Anesthesiology. 2004 Aug;101(2):461-7. doi: 10.1097/00000542-200408000-00028. PMID 15277930
- [Background] Vranceanu AM, Jupiter JB, Mudgal CS, Ring D. Predictors of pain intensity and disability after minor hand surgery. J Hand Surg Am. 2010 Jun;35(6):956-60. doi: 10.1016/j.jhsa.2010.02.001. Epub 2010 Apr 9. PMID 20381981
- Available data/document: Study Protocol: HS-15-00706 — http://istar.usc.edu
- Available data/document: Informed Consent Form: HS-15-00706 — http://istar.usc.edu